CLINICAL TRIAL: NCT03995251
Title: Efficacy and Safety of Testosterone Therapy in Improving Sarcopenia in Men With Cirrhosis a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Testosterone Therapy in Improving Sarcopenia in Men With Cirrhosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-21
Record Dates: First submitted 2019-06-19; First posted 2019-06-24 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-06

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Medical Treatment +Intramuscular Testosterone + Exerc (Experimental): Intramuscular Testosterone Undecanoate 1000 Mg (4 ml volume in oily base) will be injected into the upper, outer quadrant of the buttock at 0, 6, 12,16,20, 24 weeks according to manufacturer recommendations
  Interventions: Drug: Testosterone Supplementation; Drug: Standard Medical Treatment; Other: Exercise
- Standard Medical Treatment+Exercise (Active Comparator): Standard Medical Treatment +Exercise
  Interventions: Drug: Standard Medical Treatment; Other: Exercise

INTERVENTIONS:
Drug: Testosterone Supplementation — Intramuscular Testosterone Undecanoate 1000 Mg (4 ml volume in oily base) will be injected into the upper, outer quadrant of the buttock at 0, 6, 12,16,20, 24 weeks according to manufacturer recommendations
  Arms: Standard Medical Treatment +Intramuscular Testosterone + Exerc
Drug: Standard Medical Treatment — Standard Medical Treatment
Other: Exercise — Exercise

SUMMARY:
* Study Population- Patient with cirrhosis with any aetiology with sarcopenia visiting ILBS OPD/IPDs who are willing to visit ILBS gymnasium twice weekly for first month.
* Study Design- A Prospective Randomized Controlled Trial
* Study Period- Study will be conducted at ILBS from April 2019 to Oct 2019

  * Sample Size:As shown by Eva Roman et al - in cirhotics with sarcopenia exercise increases mean lean appendicular mass , by 0.38 kg (14 patients, p < 0.03), and Sinclair et al has shown testosterone (22 patients, p <0.05)) to increase mean Appendicular lean mass by +1.69 kg - for 10% increase in APLM
  * we need to enroll 40 patients in each arm, and considering a los to follow up approx.10% , will require minimum 44 patients in each arm
  * We will therefore enroll and randomize 100 patients with 50 in each arm.

Intervention - Testosterone Supplementation - Intramuscular Testosterone Undecanoate 1000 Mg (4 ml volume in oily base) will be injected into the upper, outer quadrant of the buttock at 0, 6, 12,16,20, 24 weeks according to manufacturer recommendations.

Monitoring and assessment - On every visit patient will be inquired or evaluated for side effects like local site pain or hematoma , hypertension, headache, allergic reactions, acne, nausea , mood swings, pedal edema , breast enlargement and others.

ELIGIBILITY:
Inclusion Criteria:

* Men with cirrhosis of any etiology
* Sarcopenia
* CTP 6-12

Exclusion Criteria:

* Hepatocellular carcinoma
* Other known malignancy,
* CTP > 12
* Acute liver injury
* Prostate disease,
* Known hypersensitivity to testosterone therapy,
* Polycythaemia (haematocrit >55%),
* Uncontrolled hypertension (>160/90 mmHg despite treatment),
* Uncontrolled obstructive sleep apnoea,
* Severe renal dysfunction (estimated glomerular filtration rate <30ml/min)
* Uncontrolled epilepsy, migraine, or significant cardiac insufficiency (New York Heart Association class III or IV or LVEF < 45-50%.
* CKD (Chronic Kidney Disease) - eGFR (Glomerular Filtration Rate) <60%
* Platelet count below 30,000 or taking warfarin
* Failure to give consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males only
Enrollment: 100 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Increase in Lean Appendicular Muscle Mass by more than 10% in both groups | 24 weeks

SECONDARY OUTCOMES:
Improvement by 10 % in Hand Grip strength in both groups | 24 weeks
Improvement by 10 % in6 minute walk distance in both groups | 24 weeks
Improvement by 10 % in the increased bone and muscle mass in both groups | 24 weeks
Improvement by 10 % L3 Skeletal Muscle Index in both groups. | 24 weeks
Improvement by 10 % in serum ammonia levels in both groups | 24 weeks
Improvement by 10 % in muscle fibres on Biopsy in both groups • | 24 weeks
Reduction in Myostatin level in both groups | 24 weeks
Improvement in MELD scores in both groups | 24 weeks
Decrease in mortality over 6 months in both groups | 24 weeks
Changes in HBA1C level in both groups | 24 weeks
Reduction in requirement of hospital admissions in both groups | 24 weeks
Decrease in TNF alpha levels in both groups | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided